CLINICAL TRIAL: NCT04531878
Title: Jian-She Wang of Children's Hospital of Fudan University
Brief Title: BSEP Function Rescue During Childhood Inhereditary Cholestatic Diseases
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSEP_FudanEK_001
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Hereditary Diseases; Cholestasis, Intrahepatic
Keywords: BSEP; ABCB11; biliary diversion; liver biopsy; gene
MeSH Terms: conditions — Genetic Diseases, Inborn; Cholestasis, Intrahepatic; Cholestasis, progressive familial intrahepatic 2 | interventions — 4-phenylbutyric acid; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BSEP trafficking abnormal group (Experimental): Patients with ABCB11 missense mutations that were speculated to affect the BSEP trafficking
  Interventions: Drug: 4-Phenylbutyrate

INTERVENTIONS:
Drug: 4-Phenylbutyrate — 4-phenylbutyrate therapy will be started at a daily dose of 200 mg kg/d divided in 2 oral doses of sodium phenylbutyrate (AMMONAPS, Swedish Orphan Inter AB). In order to get the best effect, the dose will be increased up to a maximum of 500 mg kg/d.
  Other Names: UDCA or biliary diversion

SUMMARY:
The purpose of the study is to improve the prognosis of inhereditary cholestasis caused by ABCB11 gene mutations by using BSEP function rescue drugs

DETAILED DESCRIPTION:
Bile acids function as detergents to aid digestion and as signaling molecules to regulate gene expression and metabolism. They are synthesized from cholesterol in the liver, secreted into bile and re -turned from chyme to liver in portal- vein blood 6-10 times per day (enterohepatic circulation. Enterohepatic circulation of bile acids involves more than 20 transporters among which bile salt export pump (BSEP), encoded by ABCB11 plays a key role. BSEP medi-ates the secretion of bile acids across the canalicular membrane of hepatocytes into bile to provide the osmotic pressure for bile flow. Mutations in ABCB11 can cause absence or dysfunction of BSEP leading to cholestasis. Bile acid accumulation in hepatocytes caused by BSEP dysfunction is associated with a range of liver dis-eases, ranging from transient neonatal cholestasis to fatal progressive familial intrahepatic cholestasis (PFIC), with jaundice, growth retardation, cirrhosis, liver failure and death. Our current indicates that more than 70% patents with ABCB11 mutations need liver-transplantation or dead during follow-up. In recent years, some targeted drugs including 4-phenylbutyrate(for patients with BSEP trafficking abnormal), ivacaftor(for patients with abnormal BSEP transport function), and gentamicin (for patients with none sense mutations) have emerged make it possible for individual targeted therapy possible.

ELIGIBILITY:
Inclusion Criteria:

* with signed informed consent form from the guardian, and the patient if applicable.
* aged from 2 month to 18 years old.
* with cholestatic disease caused by ABCB11 biallelic mutation.
* Long-term residence in China.

Exclusion Criteria:

* Currently receiving or previously received experimental drugs.
* The child is already in the stage of liver failure, or in unstable state that are not suitable for drug treatment according to the researcher's judgment: serious complications such as bleeding tendency and skin rash.
* accompany with other chronic liver disease (viral hepatitis B and C, autoimmune hepatitis, wilson disease, cystic fibrosis, primary biliary cirrhosis, biliary atresia, sclerosing cholangitis, bile acid synthesis defects, and infections, cholestasis caused by space-occupying and other reasons).
* Suffered from congenital TORCHES infection, including toxoplasma gondii, rubella virus, cytomegalovirus, herpes simplex virus, EB virus, syphilis, HIV, etc.
* With any other major medical conditions that may affect drug absorption, metabolism, or excretion based on the researcher's judgment.
* Known or suspected hypersensitivity to any experimental drugs or their indigents.
* Patients with alcohol or drug dependence.
* In receiving any investigational drugs or within 60 days before enrollment.

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-08 (Estimated); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Native liver survive time | During follow-up (about 3 years）
  Time of patient survived with native liver will be accessed.

SECONDARY OUTCOMES:
ALT(Alanine Aminotransferase) | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable. ALT would be measured.
DB(direct bilirubin) levels | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable. DB would be measured.
TB(total bilirubin) | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable. TB would be measured.
AST(Aspartate Aminotransferase) | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable. AST would be measured.
Weight | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable. The weight of the patients.
Length | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable. The length of the patients
Itching relief | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable.The itching score level will be accessed using a score ranged from 0 to 10.
Liver pathological staging | day 90, 180
  It is a repeated measurement variable.Liver pathological staging will be accessed using the Batts-Ludwig system.
Coagulation function | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable.The INR(international normalized ratio)/PT(prothrombin time) levels will be followed if with coagulation function abnormal.
Hypoglycemia | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable.The glucose wil be followed.
Hypo25-hydroxyvitamin Demia | at day 0, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable. Hypo25-hydroxyvitamin D levels will be followed.
The bile acid profiling | at day 30, 60, 90, 180, 360, 720 and 1080
  It is a repeated measurement variable. The bile acid profiling will be checked during follow-up.
Hypoproteinemia | at day 0, 7, 14, 28, 56, 90, 120, 180, 240, 300, 360, 540, 720 and 1080
  It is a repeated measurement variable. The albumin wil be followed.
Adverse events | During follow-up (about 3 years）
  It is a binary variable(1/0). If any adverse events including bleeding, fractures, tumors, and hepatic encephalopathy happended during the follow-up, the variable would be setted into "1". The incidence of each adverse events will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-She Wang, Ph.D, Study Chair — Children's hospital of Fudan Unviersity

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Targeted pharmacotherapy in ABCB11 mutation by 4-phenylbutyrate — http://www.ncbi.nlm.nih.gov/pubmed/25716872
- See also: Pharmacological premature termination codon readthrough of ABCB11 — http://www.ncbi.nlm.nih.gov/pubmed/32702170
- See also: Functional rescue of an ABCB11 mutant by ivacaftor — http://www.ncbi.nlm.nih.gov/pubmed/32433800